CLINICAL TRIAL: NCT03392415
Title: The NOrdic-Baltic Randomized Registry Study for Long-term Clinical Evaluation of Adjunction of PCI to Optimal Medical Therapy in Chronic Total Coronary Occlusion
Brief Title: The NOrdic-Baltic Randomized Registry Study for Evaluation of PCI in Chronic Total Coronary Occlusion
Acronym: NOBLE-CTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leif Thuesen (Other)
Responsible Party: Sponsor-Investigator, Leif Thuesen, Senior consultant, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: N-20170063
Record Dates: First submitted 2017-11-20; First posted 2018-01-08 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Chronic Total Occlusion of Coronary Artery; Heart Failure; Angina Pectoris
Keywords: chronic total occlusion; CTO; PCI; percutaneus coronary intervention
MeSH Terms: conditions — Heart Failure; Angina Pectoris

STUDY DESIGN:
Intervention Model Description: Randomized registry with option of crossover after 6months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial conservative treatment (Active Comparator): Optimal medical therapy and option for crossover after 6 months or fulfillment of certain conditions
  Interventions: Procedure: CTO PCI
- initial interventional treatment (Experimental): CTO PCI attempt as initial strategy with medical optimization simultaneously
  Interventions: Procedure: CTO PCI

INTERVENTIONS:
Procedure: CTO PCI — attempted percutaneous coronary intervention of the chronic total coronary occlusion

SUMMARY:
Randomized registry for the study of CTO PCI as adjunction to optimal medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥1 CTO lesion amenable to PCI.
* Stable and stabilized coronary artery disease
* Symptoms (angina pectoris or shortness of breath) and/or signs of reversible perfusion defect by SPECT, PET or MR and/or angiographic/echocardiographic indication of reversible ischemia.
* CTO lesion in a major coronary vessel supplying a significant myocardial territory (vessel diameter usually ≥3mm).

Exclusion Criteria:

* Expected survival <1 year.
* Renal failure on dialysis.
* Stable non-CTO lesions treated within one month.
* Declined informed consent.
* Regarding CMR: allergy to contrast medium, severe obesity, claustrophobia and certain metallic implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | a minimal follow-up of 6 months
  All-cause mortality after inclusion of 2000 patients
Quality of life assessment | 6 months.
  Quality of life assessment by 12-Item Short Form Survey Instrument (SF-12v2)

SECONDARY OUTCOMES:
MR perfusion | 6 months
  Reduction of inducible myocardial perfusion defect evaluated, improvement of left ventricular function and correlation of angina and perfusion defect
Echocardiography | 6 months
  evaluation of systolic and diastolic left ventricular function compared to index echocardiography before CTO PCI.

OTHER OUTCOMES:
Socio-economic | 1 year
  Socio-economic consequenses of CTO PCI. Treatment cost compared to coronary bypass surgery

CONTACTS AND LOCATIONS:
Overall Officials: Søren Pihlkjær Hjortshøj, MD, Study Chair — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christensen MK, Eftekhari A, Raungaard B, Steigen TK, Kumsaars I, Riahi S, Sogaard P, Thuesen L. Impact of Percutaneous Intervention Compared to Pharmaceutical Therapy on Complex Arrhythmias in Patients With Chronic Total Coronary Occlusion. Rationale and Design of the CTO-ARRHYTHMIA Study. Cardiovasc Revasc Med. 2023 Sep;54:69-72. doi: 10.1016/j.carrev.2023.04.001. Epub 2023 Apr 10. PMID 37117085
- [Derived] Rinfret S, Sandesara PB. Reducing Ischemia With CTO PCI: Good News, But Questions Remain. JACC Cardiovasc Interv. 2021 Jul 12;14(13):1419-1422. doi: 10.1016/j.jcin.2021.05.028. No abstract available. PMID 34238552

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT03392415/Prot_SAP_000.pdf